CLINICAL TRIAL: NCT07144202
Title: Study on the Immunity Persistence Following Immunization With Enterovirus Type 71 Vaccine, Inactivated (Human Diploid Cell)
Brief Title: Study on the Persistence of Immunity Following EV71 Vaccination
Status: Enrolling by invitation | Type: Observational
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: EV71-402
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Hand, Foot, and Mouth Disease; Hand, Foot, and Mouth Disease (HFMD)
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Placebo: Two doses of placebo at the vaccination schedule of Day 0, 28
- Vaccine: EV71 vaccine on Day 0, 28

SUMMARY:
This is a thirteen-year follow-up study conducted as an extension of a Phase III clinical trial. In this study, a sub-cohort of volunteers who was eligible for enrollment and randomly administrated either 2 dose EV71 vaccine or placebo in the phase III clinical trial was selected to evaluate the EV71 immune levels 13 years after the primary vaccination.

DETAILED DESCRIPTION:
The initial study was a randomized, double-blind, placebo-controlled phase III clinical trial conducted in children aged 6-71 months from Guilin region of Guangxi Province in 2012. A total of 12000 participants (with 1100 in the immunogenicity group) were randomized in a 1:1 ratio to receive two doses EV71 vaccine or placebo on a 0-, 28-day schedule. Besides, an extended one-year and two year follow-up of this study was completed in 2013.

In this study, immunogenicity group participants from the phase III clinical trial was chosen as the studied subjects. A retrospective survey for the enrolled subjects involved with the history of HFMD and the extra vaccination of EV71 vaccine was conducted before blood collection. 3 ml venous blood were collected from each available subject for EV71 neutralizing antibody (NAb) testing. Since the unblinding was performed after the initial study completed, this study was an open-labelled detection for the persistence of the vaccine-induced EV71 NAb.

ELIGIBILITY:
Inclusion Criteria:

* Included in the immunogenicity group of initial studyand randomly into either vaccine (fulfilled the two doses vaccination following the protocol) or placebo group.
* Volunteers and their legal guardians or appointed representatives must provide valid legal identification documents.
* Legal guardians or appointed representatives of volunteers must have the capacity to understand the informed consent document and the research process, voluntarily participate, sign the informed consent form, and be able to comply with the study's requirements.

Exclusion Criteria:

* Had history of extra EV71 vaccination.
* Previous history of hand-foot-mouth disease.
* Participating in other research.
* Subjects with a hereditary bleeding tendency or coagulopathy, or a history of bleeding disorders.
* Investigators' Discretion: The final exclusion criterion is the discretion of investigators to determine whether a subject is suitable for participation in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Immunogenicity group participants from the phase III clinical trial
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2025-08-10 (Actual); Primary Completion 2025-08-25 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity index-seropositive rates of neutralizing antibody | Year 13 after the second vaccination
  Neutralizing antibody assay will be performed using the neutralization and Microneutralization test method. Seropositive will be defined as the positive results with ties≥1:8
Immunogenicity index-geometric mean titer (GMT) of neutralizing antibody | Year 13 after the second vaccination
  Neutralizing antibody assay will be performed using the neutralization and Microneutralization test method

CONTACTS AND LOCATIONS:
Overall Officials: Teng Huang, Principal Investigator — Guangxi Zhuang Autonomous Region Center for Disease Prevention and Control
Locations (4):
- China (4):
  - Lingchuan Center for Disease Control and Prevention, Guilin, Guangxi
  - Lipu Center for Disease Control and Prevention, Guilin, Guangxi
  - Xing'an Center for Disease Control and Prevention, Guilin, Guangxi
  - Yongfu Center for Disease Control and Prevention, Guilin, Guangxi

IPD SHARING:
Plan to Share IPD: No